CLINICAL TRIAL: NCT01266044
Title: Controlled Trial Of Acupuncture To Prevent Radiation-Induced Xerostomia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-0584; NCI-2011-00306 (Registry Identifier: NCI CTRP); R01CA148707-01A1 (NIH)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Head And Neck Cancer
Keywords: Radiation-induced xerostomia; Acupuncture; Oropharyngeal cancer; Radiation Therapy; IMRT; Dry mouth
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Xerostomia | interventions — Standard of Care; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture - Group 1 (Experimental): Acupuncture at 14 points. The needles will remain in place for 20 minutes with each treatment. Questionnaires - Baseline assessments will be completed within 7 days prior to starting radiotherapy, and patients will then complete the same assessments again at week 4 and 7 of radiotherapy and 3, 6, and 12 months after the end of radiotherapy.
  Interventions: Procedure: Acupuncture - Group 1; Other: Standard Care; Other: Questionnaire
- Acupuncture - Group 2 (Active Comparator): Acupuncture needles placed at different points from Group 1. The needles will remain in place for 20 minutes with each treatment. Questionnaires - Baseline assessments will be completed within 7 days prior to starting radiotherapy, and patients will then complete the same assessments again at week 4 and 7 of radiotherapy and 3, 6, and 12 months after the end of radiotherapy.
  Interventions: Procedure: Acupuncture - Group 2; Other: Standard Care; Other: Questionnaire
- Standard Care (Other): Standard oral care recommendations. Participants in all groups will receive the same recommendations. Questionnaires - Baseline assessments will be completed within 7 days prior to starting radiotherapy, and patients will then complete the same assessments again at week 4 and 7 of radiotherapy and 3, 6, and 12 months after the end of radiotherapy.
  Interventions: Other: Standard Care; Other: Questionnaire

INTERVENTIONS:
Procedure: Acupuncture - Group 1 — Acupuncture at 14 points. The needles will remain in place for 20 minutes with each treatment.
  Arms: Acupuncture - Group 1
Procedure: Acupuncture - Group 2 — Acupuncture needles placed at different points from Group 1. The needles will remain in place for 20 minutes with each treatment.
  Arms: Acupuncture - Group 2
Other: Standard Care — Standard oral care recommendations. Participants in all groups will receive the same recommendations.
Other: Questionnaire — Baseline assessments will be completed within 7 days prior to starting radiotherapy, and patients will then complete the same assessments again at week 4 and 7 of radiotherapy and 3, 6, and 12 months after the end of radiotherapy.

SUMMARY:
The goal of this clinical research study is to learn if acupuncture can help to prevent xerostomia (dry mouth) and improve the quality of life in patients who receive radiation treatment to the head and neck. This study will determine if one acupuncture treatment approach is more effective than another. Dry mouth is a common problem among cancer patients who have received radiation treatment to the head and neck.

DETAILED DESCRIPTION:
Acupuncture is a technique that may treat symptoms by inserting very thin, solid, sterile, stainless steel needles into the skin at specific points.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of a dice) into 1 of 3 groups.

Group 1 will receive acupuncture during the radiation treatment period.

Group 2 will receive acupuncture at different points on the body than those in Group 1 during the radiation treatment period.

You will not know if you are assigned to Group 1 or 2.

Group 3 will receive standard care without any kind of acupuncture during the radiation treatment period.

Study Visits:

If you are in Group 1 and 2, you will receive up to 21 acupuncture treatments with no more than 3 treatments per week during your regularly scheduled radiotherapy visits. It will take about 20 minutes to complete the acupuncture session each time.

No matter which group you are assigned to, you will complete the following at the middle and end of radiotherapy treatment, and again 2-4, 5-9, 10-15 months after radiotherapy treatment is complete:

* Your vital signs will be recorded.
* You will be asked about any drugs you are taking.
* You will complete 9 questionnaires about your dry mouth, quality of life, and mood. It should take about 30 minutes in total to complete the questionnaires. If you are not able to complete the questionnaires during your regularly scheduled visits, you will be able to take the questionnaires home to complete them and will be given a postage-paid return envelope to mail them back to the study doctor.
* A saliva sample will be collected to measure the quality and amount of saliva produced during radiotherapy.
* You will complete a form about your oral hygiene that should take about 5 minutes to complete.

Length of Study:

You will remain on study for up to 17 months.

Additional Information:

After your participation on this study is complete and you are no longer enrolled in this study, if you were in Group 2 or 3, you will be offered to receive 3 acupuncture treatments.

This is an investigational study.

Up to 435 patients will take part in this multicenter study. Up to 193 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and be able to give informed consent.
2. Diagnosed with head and neck cancer, which will be primarily oropharyngeal, and scheduled to undergo IMRT with or without concurrent chemotherapy at M. D. Anderson.
3. Treatment plan that includes external beam radiation at a mean dose of at least 24 Gy or more to one of the parotid glands (the other gland can receive less than 24 Gy).
4. Anatomically intact parotid and submandibular glands.
5. Karnofsky performance status > 60.

Exclusion Criteria:

1. History of xerostomia prior to head and neck radiation therapy or history of Sjögren's disease or another underlying systemic illness known to cause xerostomia.
2. Prior head and neck radiation treatment.
3. Suspected or confirmed physical closure of salivary gland ducts on either side.
4. Known bleeding disorders or taking any dose of warfarin or heparin.
5. Upper or lower extremity deformities that could interfere with accurate acupoint location or alter the energy pathway as defined by traditional acupuncture theory.
6. Local skin infections at or near the acupuncture sites or active systemic infection.
7. History of cerebrovascular accident or spinal cord injury since the mechanism of acupuncture may be associated with central nervous system activity.
8. Mental incapacitation or significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry as these patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.
9. Current acknowledged use of any illicit drugs or evidence of alcohol abuse as defined by The American Psychiatric Association criteria.
10. Current acknowledged use of amifostine, cholinergic agonist medications (pilocarpine, cevimeline), certain beta adrenergic antagonists, anticholinergic agents, or any saliva substitute or other medication/herbal preparation known to affect salivary function (see Appendix F).
11. Patients who are currently receiving acupuncture for any condition or if they have ever had acupuncture before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2011-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Xerostomia Symptoms Using the Xerostomia Questionnaire (XQ) | 4 weeks
  Xerostomia Questionnaire (XQ), an 8-item questionnaire where subjects rate each symptom on an 11-point ordinal Likert scale from 0 to 10, with higher scores indicating greater dryness or discomfort due to dryness.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Garcia MK, Meng Z, Rosenthal DI, Shen Y, Chambers M, Yang P, Wei Q, Hu C, Wu C, Bei W, Prinsloo S, Chiang J, Lopez G, Cohen L. Effect of True and Sham Acupuncture on Radiation-Induced Xerostomia Among Patients With Head and Neck Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1916910. doi: 10.1001/jamanetworkopen.2019.16910. PMID 31808921
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org